CLINICAL TRIAL: NCT05216263
Title: A Phase 3 Multicenter 24-Week Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Atogepant When Added to OnabotulinumtoxinA (BOTOX) for the Preventive Treatment of Chronic Migraine
Brief Title: Study of Oral Atogepant When Added to OnabotulinumtoxinA (BOTOX) to Assess Adverse Events and Change in Disease Activity in Adult Participants With Chronic Migraine
Acronym: ATO-BOTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22-418
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; Migraine; Atogepant; OnabotulinumtoxinA; BOTOX; QULIPTA
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atogepant (Experimental): Participants will receive atogepant once a day (QD) during the 24-week treatment period.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: QULIPTA

SUMMARY:
Migraine is characterized by attacks of throbbing, moderate or severe headache, often associated with nausea, vomiting, and/or sensitivity to light and/or sound. The study will assess safety and tolerability of atogepant when added to BOTOX, as well as prospectively evaluate the efficacy of add-on atogepant for migraine prevention. Adverse events and change in disease activity will be monitored.

Atogepant is an investigational drug being developed to prevent chronic migraine. Approximately 75 adult participants will be enrolled at approximately 30 sites in the United States.

All participants will receive atogepant oral tablet once a day (QD) during the 24-week treatment period, in addition to their standard of care Botox.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of chronic migraine (CM), with or without aura, consistent with a diagnosis according to International Classification of Headache Disorders 3rd edition (ICHD-3 2018) and with or without acute medication overuse as defined in the protocol.
* Must be currently treated with BOTOX for CM: treated with >= 2 treatment cycles in the 8 months prior to Visit 2 (Day 1) with documentation of payer authorization or written attestation of self-pay to support continued use of BOTOX.
* Must have 8 to 23 (inclusive) migraine days in the electronic diary [eDiary] screening/baseline period (eDiary data must have been collected for at least 20 days).

Exclusion Criteria:

* Use of opioid-containing products for more than 4 days per month for acute treatment of headache in the 3 months prior to Screening or during the screening/baseline period.
* Treatment of study target muscles using acupuncture, transcutaneous electrical nerve stimulation (TENS), cranial traction, dental splints for headache, or head and/or neck injections of anesthetics/steroids within 4 weeks prior to Screening and throughout the study.
* Concurrent use of any migraine prevention treatment other than BOTOX (required concomitant medication; or topiramate <=100mg daily) including use of oral gepants in the 4 weeks prior to screening nor during the screening/baseline period.
* Current use or use within the 6 months (24 weeks) prior to Screening, of mAbs blocking the CGRP pathway.
* Concurrent use of oral gepants for acute migraine treatment in the 4 weeks prior to screening nor during the screening/baseline period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately 28 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Responder Status of at least 25% Reduction in the Frequency of Monthly Migraine Days Collected via Daily Electronic Diary (eDiary) | Baseline (Week 0) through 24 Weeks
  Percentage of participants achieving at least 25% reduction from baseline in the frequency of monthly migraine days will be assessed.
Responder Status of at least 30% Reduction in the Frequency of Monthly Migraine Days Collected via eDiary | Baseline (Week 0) through 24 Weeks
  Percentage of participants achieving at least 30% reduction from baseline in the frequency of monthly migraine days will be assessed.
Responder Status of at least 50% Reduction in the Frequency of Monthly Migraine Days Collected via eDiary | Baseline (Week 0) through 24 Weeks
  Percentage of participants achieving at least 50% reduction from baseline in the frequency of monthly migraine days will be assessed.
Responder Status of at least 75% Reduction in the Frequency of Monthly Migraine Days Collected via eDiary | Baseline (Week 0) through 24 Weeks
  Percentage of participants achieving at least 75% reduction from baseline in the frequency of monthly migraine days will be assessed.
Responder Status of at least 100% Reduction in the Frequency of Monthly Migraine Days Collected via eDiary | Baseline (Week 0) through 24 Weeks
  Percentage of participants achieving at least 100% reduction from baseline in the frequency of monthly migraine days will be assessed.
Change From Baseline in Monthly Migraine Days | Baseline (Week 0) through 24 Weeks
  Change from Baseline in monthly migraine days, defined by International Headache Society (IHS) Guidelines 2018 will be assessed.
Change from Baseline in Monthly Headache Days, Moderate or Severe Headache Days, Cumulative Hours of Headache, Acute Treatment Medication Use Days, Headache Free Days, and Migraine Symptom-Free Days | Baseline (Week 0) through 24 Weeks
  Change from baseline in monthly headache days, moderate or severe headache days, cumulative hours of headache, acute treatment medication use days, headache free days, and migraine symptom-free days, defined by IHS Guidelines 2018 will be assessed.
Change from Baseline in Monthly days with Non-Headache Migraine Symptoms | Baseline (Week 0) through 24 Weeks
  Change from baseline in monthly days with non-headache migraine symptoms such as photophobia, phonophobia, nausea and/or vomiting, dizziness, neck pain, tiredness, mood change, yawning, thirst, cravings, urinary frequency, cranial autonomic symptoms
Change from Baseline in Monthly Activity Impairment in Migraine - Diary (AIM-D) | Baseline (Week 0) through 24 Weeks
  The AIM-D is an 11-item daily diary measure that assesses the impact of migraine and is comprised of two domains that evaluate performance of daily activities (7 items) and physical impairment (4 items).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (29):
- United States (29):
  - Neurology and Neurodiagnostics of Alabama /ID# 242538, Hoover, Alabama
  - Barrow Neurological Institute - Dignity Health St. Joseph's Hosp and Medical Ctr /ID# 241812, Phoenix, Arizona
  - Arkansas Clinical Research /ID# 241789, Little Rock, Arkansas
  - Hope Clinical Research /ID# 241772, Canoga Park, California
  - Profound Research LLC /ID# 244084, Carlsbad, California
  - Neuro Pain Medical Center /ID# 241992, Fresno, California
  - Neurological Research Institute /ID# 242688, Santa Monica, California
  - Neurology Offices of South Florida, PLLC /ID# 242693, Boca Raton, Florida
  - Coastal Clinical Research Specialists /ID# 247992, Jacksonville Beach, Florida
  - University of Miami /ID# 252230, Miami, Florida
  - First Physicians Group - Waldemere /ID# 242861, Sarasota, Florida
  - Kansas Institute of Research /ID# 241796, Overland Park, Kansas
  - Ochsner Clinic Foundation /ID# 241803, Covington, Louisiana
  - Beth Israel Deaconess Medical Center /ID# 241800, Boston, Massachusetts
  - Michigan Headache & Neurological Institute (MHNI) /ID# 241784, Ann Arbor, Michigan
  - Minneapolis Clinic of Neurology - Burnsville /ID# 241994, Burnsville, Minnesota
  - Albany Medical College /ID# 242757, Albany, New York
  - Dent Neurologic Institute - Amherst /ID# 241776, Amherst, New York
  - Headache Wellness Center /ID# 241791, Greensboro, North Carolina
  - Jefferson Hospital for Neuroscience /ID# 243712, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians - Jacob Murphy /ID# 241798, Uniontown, Pennsylvania
  - Chattanooga Medical Research /ID# 253295, Chattanooga, Tennessee
  - Nashville Neuroscience Group /ID# 243592, Nashville, Tennessee
  - Texas Neurology /ID# 241795, Dallas, Texas
  - Inova Health System /ID# 252242, Falls Church, Virginia
  - Integrated Neurology Services - Falls Church /ID# 244747, Falls Church, Virginia
  - Puget Sound Neurology /ID# 241787, Tacoma, Washington
  - Frontier Clinical Research - Kingwood /ID# 242928, Kingwood, West Virginia
  - West Virginia Univ School Med /ID# 252869, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-418